CLINICAL TRIAL: NCT05009329
Title: Multi-center, Open, Dose-escalation, and Expanded Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of JAB-21822 in Advanced Solid Tumors With KRAS p.G12C Mutation
Brief Title: A Study of JAB-21822 in Adult Patients With Advanced Solid Tumors Harboring KRAS p.G12C Mutation in China
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-1002
Record Dates: First submitted 2021-07-26; First posted 2021-08-17 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: NSCLC; Solid Tumor
Keywords: KRAS p.G12C Mutant Advanced Solid Tumor; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1 Dose Exploration (Experimental): Dose escalation of JAB-21822 to determine maximum tolerated dose.
  Interventions: Drug: JAB-21822
- Phase IIa Dose Expansion (Experimental): Patients with KRAS p.G12C mutant advanced non small cell lung cancer or other solid tumors will be enrolled and treated at the monotherapy RP2D to evaluate the safety and preliminary efficacy.
  Interventions: Drug: JAB-21822
- Phase IIb (Experimental): Patients with KRAS p.G12C mutant advanced non small cell lung cancer will be enrolled and treated at the monotherapy RP2D to evaluate the safety and efficacy.
  Interventions: Drug: JAB-21822

INTERVENTIONS:
Drug: JAB-21822 — JAB-21822 will be administered orally
  Other Names: glecirasib
  Arms: Phase 1 Dose Exploration
Drug: JAB-21822 — JAB-21822 will be administered orally
  Other Names: glecirasib
  Arms: Phase IIa Dose Expansion
Drug: JAB-21822 — JAB-21822 will be administered orally
  Other Names: glecirasib
  Arms: Phase IIb

SUMMARY:
To assess safety, tolerability, PK, efficacy and determine recommended phase 2 dose (RP2D) of JAB-21822 (glecirasib) administered in adult participants with KRAS p.G12C-mutant advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Advanced (metastatic or unresectable) KRAS p.G12C mutant solid tumors, with failure or absence of standard treatment
3. Subject must be ≥18 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
5. Subjects with life expectancy ≥3 months.
6. Subjects must have at least one measurable lesion as defined by RECIST v1.1.
7. There was no serious organ dysfunction in the screening stage
8. Male or female subjects of reproductive age agree to use adequate contraception

Exclusion Criteria:

1. History of intestinal disease or major gastric surgery or inability to swallow oral medications
2. Other active cancer
3. Previously treated with KRAS G12C inhibitor
4. Active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
5. Impaired heart function or clinically significant heart disease
6. Pregnant or breast-feeding
7. Previous allogeneic bone marrow transplant or organ transplant
8. Intended study subjects who were unable to abstain from alcohol during medication
9. Other unqualified conditions judged by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) in the dose escalation phase | first 21 days
  Number of participants with dose limiting toxicities
Number of participants with adverse events | up to 3 years
  Patients will be assessed for incidence and severity of adverse events (AEs) according to NCI-CTCAE criteria
Overall response rate (ORR) by IRC (independent review committee) | up to 3 years
  ORR is defined as the proportion of participants with complete response and partial response (CR+PR) per RECIST v 1.1

SECONDARY OUTCOMES:
Overall response rate (ORR) by investigator | up to 3 years
  ORR is defined as the proportion of participants with complete response and partial response (CR+PR) per RECIST v 1.1
Duration of response ( DOR ) | up to 3 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Disease Control Rate ( DCR ) | up to 3 years
  DCR is defined as percentage of participants with complete response (CR), partial response (PR), and stable disease(SD) per RECIST v1.1
Progression-free survival (PFS) | up to 3 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death per RECIST v1.1, which occurs first
Time to response (TTR) | up to 3 years
  Time from patient randomization (first treatment) to first response per RECIST 1.1 criteria
Peak Plasma Concentration (Cmax) | up to 3 years
  Cmax of JAB-21822 will be measured by using plasma PK samples

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Wang Z, Huang J, Ba Y, Cao B, Luo S, Li W, Bai C, Song Z, Xiong J, Zhu L, An G, Zhang Y, Li Z, Li Y, Gu Y, Hu C, Li X, Huang C, Fu Q, Yin X, Liang X, Zhong D, Shi H, Li X, Li Z, Liu L, Wang F, Liang R, Xia G, Wang Z, Wang-Gillam A, Ding Y, Rao Z, Pan W, Lu S, Sun X, Shen L. Glecirasib with or without cetuximab in previously treated locally advanced or metastatic colorectal cancer with KRASG12C mutation (JAB-21822-1002 and JAB-21822-1007): two open-label, non-randomised phase 1/2 trials. Lancet Gastroenterol Hepatol. 2026 Feb;11(2):110-123. doi: 10.1016/S2468-1253(25)00267-5. Epub 2025 Dec 1. PMID 41344351
- [Derived] Li J, Deng T, Gu Y, Calles Blanco A, Li Z, Bai C, Wu L, Huang J, Li X, Yao Y, Song Z, Li Y, Liu L, Xing L, Wu W, Martinez-Perez J, Hubert A, Zugazagoitia J, Zhang J, Wang Y, Zhao Y, Wen G, Xia G, Zhong D, Chen X, Jiang K, Wang-Gillam A, Ding Y, Liu S, Rao Z, Liu X, Shen L. Efficacy and safety of glecirasib in solid tumors with KRAS G12C mutation: A pooled analysis of two phase I/II trials. Cancer Commun (Lond). 2025 Nov;45(11):1500-1512. doi: 10.1002/cac2.70056. Epub 2025 Oct 2. PMID 41037823
- [Derived] Shi Y, Fang J, Xing L, Yao Y, Zhang J, Liu L, Wang Y, Hu C, Xiong J, Liu Z, Yang R, Wang Z, Zhao E, Wang M, Zhao Y, Tang K, Li Z, Song Z, Li Y, Zhuang W, Jin B, Cheng Y, Hu Y, Gu Y, Wu L, Ma R, Yu Q, Yu Y, Zhao J, Zhao H, Lv D, Shang Y, Xing P, Zhou J, Li X, Liu Z, Dai Z, Xia G, Chen X, Ba Y, Bai C, Li Q, An G, Hu W, Wang Y, Wang-Gillam A, Ding Y, Li Q, Rao Z. Glecirasib in KRASG12C-mutated nonsmall-cell lung cancer: a phase 2b trial. Nat Med. 2025 Mar;31(3):894-900. doi: 10.1038/s41591-024-03401-z. Epub 2025 Jan 6. PMID 39762419